CLINICAL TRIAL: NCT00235846
Title: Endoscopic Vessel Harvesting During Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jan Jesper Andreasen, MD, PhD, Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VN 2004/14
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Arteriosclerosis
Keywords: Endoscopic vein harvesting; Saphenous vein
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional vein harvest (Active Comparator): Conventional open vein harvest from the lower leg
  Interventions: Procedure: vein harvest
- Endoscopic vein harvest (Experimental): Endoscopic vein harvest from the calf
  Interventions: Procedure: vein harvest

INTERVENTIONS:
Procedure: vein harvest — Conventional open vein harvest or endoscopic vein harvest

SUMMARY:
Conventional open vein harvesting from the legs during coronary artery bypass surgery result in wound complications among 30% of the patients. Endoscopic harvesting decrease the complication rate, but it remains to be shown whether this is also a fact among patient in whom only short segments of veingraft material is needed from the leg. We hypothesise that the rate of wound complications will be reduced and the patient satisfaction will be increased also among patients in whom only short vein segments are endoscopically harvested compared to conventional open vein harvesting.

DETAILED DESCRIPTION:
Conventional open vein harvesting from the legs during coronary artery bypass surgery result in wound complications among 30% of the patients. Endoscopic harvesting decrease the complication rate, but it remains to be shown whether this is also a fact among patient in whom only short segments of veingraft material is needed from the leg. We hypothesise that the rate of wound complications will be reduced and the patient satisfaction will be increased also among patients in whom only short vein segments are endoscopically harvested compared to conventional open vein harvesting.

Preoperative demographic as well ass peri- and postoperative data are collected prospectively at 5-7 days and 1 month postoperatively. Wound complications are registered as well as post operative pain in the wound is evaluated using af visual analogue scale. Patients are evaluating the cosmetic results after wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass surgery

Exclusion Criteria:

* Leg wounds
* Acute surgery
* Previous vascular surgery
* Combined surgery (valve + coronary)
* Arterial revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Rate of wound complications | 30 days
Patient satisfaction | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Andreasen, MD, Principal Investigator — Department of Cardiothoracic Surgery, Aalborg hospital, Hobrovej, postboks 365, DK-9100 Aalborg, Denmark
Locations (1):
- Aalborg Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Andreasen JJ, Nekrasas V, Dethlefsen C. Endoscopic vs open saphenous vein harvest for coronary artery bypass grafting: a prospective randomized trial. Eur J Cardiothorac Surg. 2008 Aug;34(2):384-9. doi: 10.1016/j.ejcts.2008.04.028. Epub 2008 May 27. PMID 18508277